CLINICAL TRIAL: NCT03386825
Title: COLONG: Metastatic Colorectal Cancer Patients With Long-term Response to Regorafenib
Brief Title: Metastatic Colorectal Cancer Patients With Long-term Response to Regorafenib
Acronym: COLONG
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19577
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Regorafenib_DoT<4 months: DoT < 4 months
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Regorafenib_4 months ≤ DoT < 12 months: 4 months ≤ DoT < 12 months
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)
- Regorafenib_DoT ≥ 12 months: DoT ≥ 12 months
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Antineoplastic agents, protein kinase inhibitor (L01XE21)

SUMMARY:
The aim of this local NIS(Non-Interventional Study) is to determine the proportion of Belgian patients with a duration of treatment(DoT) to Stivarga of 4 months or more in relation to the total population of Belgian metastatic colorectal cancer(mCRC) patients who were treated with Stivarga between the 1st of July 2015 and 31 July 2017. In addition, this study aims to describe the clinical characteristics of Belgian patients with a short- or long-term DoT to Stivarga.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age.
* Patients who suffer from mCRC and who started treatment with Stivarga between the 1st of July 2015 and 31 July 2017.
* Patients who already received alternative treatment options before Stivarga for the treatment of mCRC or who were not eligible for other treatment options.
* Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1 at start of Stivarga treatment.
* Sufficient kidney, liver and bone marrow function start of Stivarga treatment.
* Life expectancy ≥ 3 months at start of Stivarga treatment

Exclusion Criteria:

- Patients participating in an investigational program/clinical trial with interventions outside of routine clinical practice during the observational period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Belgian mCRC patients who were treated with Stivarga between the 1st of July 2015 and 31 July 2017.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a DoT to Stivarga of more than 4 months versus total study sample | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
ECOG performance status (0, 1) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  ECOG: Eastern Cooperative Oncology Group
Primary site of disease | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  Rectum, Left-sided colon, Right-sided colon, Colon and rectum, Transverse, Unknown (in colon)
Tumor resection (yes, no, unknown) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
Specific site of metastasis | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  Lung, Liver, Bone, Extraregional nodes, Peritoneum, Multiple, Unknown
KRAS mutation (yes, no, unknown) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
RAS mutation (yes, no, unknown) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
BRAF mutation (yes, no, unknown) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017

SECONDARY OUTCOMES:
Start date of Stivarga treatment | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
Number of prior treatment lines for metastatic cancer larger than 3 (yes, no, unknown) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
Reason for discontinuation of Stivarga treatment | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  progression - symptomatic, Progression - radiological, Progression - radiological + symptomatic, Progression - unknown, Intolerability, Death, other, unknown, not applicable
Subsequent mCRC treatment | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  Chemotherapy IV, Chemotherapy oral, Biologic therapy, Chemotherapy + biologic therapy, BSC, Other, Unknown, Not applicable
Last daily Stivarga dose | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017
  80 mg, 120 mg, 160 mg, other, unknown
Duration of treatment (months) | Retrospective chart review from 1-Jul-2015 to 1-Dec-2017

CONTACTS AND LOCATIONS:
Locations (1):
- Belgium, Multiple Locations, Belgium